CLINICAL TRIAL: NCT03925233
Title: Sensitivity Detection and Drug Resistance Mechanism of Breast Cancer Therapeutic Drugs Based on Organ-like Culture
Brief Title: Breast Cancer Treatment Based on Organ-like Culture
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY20182079-F-1
Record Dates: First submitted 2019-03-30; First posted 2019-04-24 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-03

CONDITIONS: Breast Cancer Organoids
Keywords: Drug sensitivity experiment; Resistance mechanism research
MeSH Terms: interventions — Trastuzumab; Doxorubicin; Epirubicin; Fluorouracil; Paclitaxel; Gemcitabine; Cisplatin; Endostatins; pirarubicin; pyrrolidine; ixabepilone; Tamoxifen; Vinorelbine; Carboplatin; Methotrexate; eribulin; Toremifene; Anastrozole; Letrozole; exemestane; Fulvestrant; olaparib; Bevacizumab; apatinib; Capecitabine; Cyclophosphamide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HER2+ Breast Cancer
  Interventions: Drug: Trastuzumab; Drug: Doxorubicin Hydrochloride; Drug: Epirubicin hydrochloride; Drug: Fluorouracil; Drug: Paclitaxel; Drug: Gemcitabine; Drug: Cisplatin; Drug: Recombinant Human Endostatin; Drug: Pirarubicin hydrochloride; Drug: Pyrrolidine; Drug: Ixabepilone; Drug: Tamoxifen citrate; Drug: Vinorelbine tartrate; Drug: Carboplatin; Drug: Methotrexate; Drug: Eribulin mesylate; Drug: Toremifene citrate; Drug: Anastrozole; Drug: Letrozole; Drug: Exemestane; Drug: Fulvestrant; Drug: Olaparib; Drug: Bevacizumab; Drug: Apatinib mesylate; Drug: Pattozumab; Drug: Capecitabine; Drug: Ear particles; Drug: Aidi Injection; Drug: Cyclophosphamide
- ER+ Breast Cancer
  Interventions: Drug: Trastuzumab; Drug: Doxorubicin Hydrochloride; Drug: Epirubicin hydrochloride; Drug: Fluorouracil; Drug: Paclitaxel; Drug: Gemcitabine; Drug: Cisplatin; Drug: Recombinant Human Endostatin; Drug: Pirarubicin hydrochloride; Drug: Pyrrolidine; Drug: Ixabepilone; Drug: Tamoxifen citrate; Drug: Vinorelbine tartrate; Drug: Carboplatin; Drug: Methotrexate; Drug: Eribulin mesylate; Drug: Toremifene citrate; Drug: Anastrozole; Drug: Letrozole; Drug: Exemestane; Drug: Fulvestrant; Drug: Olaparib; Drug: Bevacizumab; Drug: Apatinib mesylate; Drug: Pattozumab; Drug: Capecitabine; Drug: Ear particles; Drug: Aidi Injection; Drug: Cyclophosphamide
- Triple Negative Breast Cancer
  Interventions: Drug: Trastuzumab; Drug: Doxorubicin Hydrochloride; Drug: Epirubicin hydrochloride; Drug: Fluorouracil; Drug: Paclitaxel; Drug: Gemcitabine; Drug: Cisplatin; Drug: Recombinant Human Endostatin; Drug: Pirarubicin hydrochloride; Drug: Pyrrolidine; Drug: Ixabepilone; Drug: Tamoxifen citrate; Drug: Vinorelbine tartrate; Drug: Carboplatin; Drug: Methotrexate; Drug: Eribulin mesylate; Drug: Toremifene citrate; Drug: Anastrozole; Drug: Letrozole; Drug: Exemestane; Drug: Fulvestrant; Drug: Olaparib; Drug: Bevacizumab; Drug: Apatinib mesylate; Drug: Pattozumab; Drug: Capecitabine; Drug: Ear particles; Drug: Aidi Injection; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Trastuzumab — Trastuzumab Injection
Drug: Doxorubicin Hydrochloride — Doxorubicin Hydrochloride Injection
Drug: Epirubicin hydrochloride — Epirubicin hydrochloride injection
Drug: Fluorouracil — Fluorouracil injection
Drug: Paclitaxel — Paclitaxel injection
Drug: Gemcitabine — Gemcitabine injection
Drug: Cisplatin — Cisplatin injection
Drug: Recombinant Human Endostatin — Recombinant Human Endostatin Injection
Drug: Pirarubicin hydrochloride — Pirarubicin hydrochloride injection
Drug: Pyrrolidine — Pyrrolidine tablets
Drug: Ixabepilone — Ixapilone Injection
Drug: Tamoxifen citrate — Tamoxifen citrate tablets
Drug: Vinorelbine tartrate — Vinorelbine tartrate injection
Drug: Carboplatin — Carboplatin injection
Drug: Methotrexate — Methotrexate injection
Drug: Eribulin mesylate — Eribulin mesylate injection
Drug: Toremifene citrate — Toremifene citrate tablets
Drug: Anastrozole — Anastrozole tablets
Drug: Letrozole — Letrozole tablets
Drug: Exemestane — Exemestane tablets
Drug: Fulvestrant — Fulvestrant injection
Drug: Olaparib — Olapani pill
Drug: Bevacizumab — Bevacizumab injection
Drug: Apatinib mesylate — Apatinib mesylate tablets
Drug: Pattozumab — Pattozumab injection
Drug: Capecitabine — Capecitabine tablets
Drug: Ear particles — Ear particles
Drug: Aidi Injection — Aidi Injection
Drug: Cyclophosphamide — Cyclophosphamide injection

SUMMARY:
Based on the breast cancer organ platform, this experiment establishes a drug sensitivity test method that is closer to the body tumor in breast cancer, provides a basis for the accurate treatment of breast cancer, and discusses the possible mechanism of breast cancer drug resistance.

ELIGIBILITY:
Inclusion Criteria:

Patients with breast cancer and the largest tumor diameter ≥ 3cm No previous chemotherapy regimen age 18-65 years old Can obtain the tumor tissue specimens required for culture Heart, liver, kidney and bone marrow hematopoietic function is good Know and sign the informed consent form

Exclusion Criteria:

Pregnant or lactating women Also suffering from other cancer patients There are serious uncontrolled medical diseases or acute infections Those who are known to be allergic to this study drug or a variety of previous drugs The patient cannot understand the purpose of the study or disagree with the requirements of the study.

Other investigators believe that patients who are not suitable for this study group

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: With the prolongation of human life and lifestyle changes, the incidence and mortality of cancer has increased year by year. Since 2010, cancer has become the leading cause of death. Among women, the incidence of breast cancer is the highest, and it shows a growing trend, which seriously threatens women's health. Breast cancer has a high degree of tumor heterogeneity, which leads to a great difference in sensitivity to chemotherapy among affected individuals. The drug resistance after chemotherapy leads to poor prognosis. Therefore, screening for breast cancer tumor cells is sensitive to chemotherapy. Molecular level studies of drug resistance are necessary.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-01-02 (Actual); Primary Completion 2021-12-15 (Estimated); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
Detection of cell viability | 8 weeks before neoadjuvant chemotherapy
  1. The organ-like organ was assayed for cell viability using CellTiter Glo 3D reagent, and the curve was used to obtain a half-inhibitory concentration range. The dose was adjusted according to the half-inhibition concentration range to obtain an accurate half-inhibitory concentration.

SECONDARY OUTCOMES:
Detection of in vitro model drug sensitivity | 8 weeks before neoadjuvant chemotherapy
  2. In vitro model drug sensitivity: sensitive and insensitive
Clinical efficacy assessment according to RECIST criteria | 8 weeks before neoadjuvant chemotherapy
  Clinical efficacy evaluation according to RECIST criteria: imaging ultrasonography, histological pathology.

CONTACTS AND LOCATIONS:
Locations (1):
- JingSu, Xi'an, Shaanxi, China